Version no. 2 08/08/2022

| Identification number: |
|------------------------|

## THE CHINESE UNIVERSITY OF HONG KONG

## Survey and Behavioural Research Ethics

## **Information sheet and Consent Form**

#### **Information sheet**

# Study Title:

The effectiveness of an educational program on the mental health literacy of nurses working in general hospitals: a controlled trial

# Name of the Principal Investigator:

Ms. CHEUNG, Janice (Student of Doctor of Nursing, The Chinese University of Hong Kong)

# Name of research supervisor:

Professor Cheng, Ho Yu (The Nethersole School of Nursing, The Chinese University of Hong Kong)

## Department:

The Nethersole School of Nursing, Faculty of Medicine, The Chinese University of Hong Kong

Castle Peak Hospital, Department of General Adult Psychiatry, New Territories West Cluster, Hospital Authority

You are invited to participate in this research study. Please read the information carefully and take time to decide whether you wish to participate in the study.

Version no. 2 08/08/2022

# **Description of the study:**

This study aims to examine the effect of an educational program (Mental Health Literacy Program) on improving the mental health literacy of general hospital nurses, in terms of knowledge of mental health, mental problems, or their treatment; attitude, or stigma about mental problems; and help-seeking efficacy. It also measures the interventional effect on perceived competency in caring for patients with mental illness and work stress among general hospital nurses, as well as patient satisfaction with nursing care in general hospitals. Your participation will take 11 weeks.

### Method:

Participants will be assigned to either an intervention group or a control group. Intervention group: You will receive a Mental Health Literacy Program consisting of six 30-minutes online educational sessions and one 60-minutes face-to-face session. Control group: No active intervention.

All participants (intervention and control groups) will be asked to complete sets of questionnaires regarding the level of mental health literacy, perceived competency in caring for patients with mental illnesses, and the work stress level at baseline, 7 weeks, and 11 weeks after joining the study. The time for completion of the questionnaire should take about 15 minutes.

**Target participants:** Full time registered nurse (general) or enrolled nurse (general) who provides care to adult patients in emergency departments or medical wards, can communicate and understand Chinese and English, and have access to the internet.

**Risks:** There is no risk of physical or mental harm for participating in this study.

**Benefits:** The findings of this study are expected to provide evidence-based data on the application of the educational program in healthcare organizations to improve the mental health literacy of nurses working in general hospitals. New knowledge can be generated, which can aid in the development of an in-service training program targeted at improving clinical practices for patients with mental illnesses in general hospitals.

**Compensation:** a cash coupon of HKD 50 will be given to the participant who completes all the measurements to compensate for the time spent.

**Information protection:** Any information obtained in connection with this study will remain confidential and at no time will your name be identified in any report of this

study. In any writing or presentations, we will use a made-up name for you. No one except investigators will know about your specific answers. Your identity will be removed from all records after the study. Only the research team, New Territories East Cluster Clinical Research Ethics Committee (NTEC REC), and New Territories West Cluster Research Ethics Committee (NTWC REC) access the subject's record related to the study for research and ethics review purposes.

**Voluntary participation:** Please understand that your participation is voluntary, and you are free to withdraw from the study and discontinue participation at any time without any consequences.

Contact details: If you have any questions about participation in this study, you may contact Ms. CHEUNG, Janice at <a href="mailto:1155149877@link.cuhk.edu.hk">1155149877@link.cuhk.edu.hk</a> or research supervisor Dr. Cheng, H.Y. at <a href="mailto:hycheng@cuhk.edu.hk">hycheng@cuhk.edu.hk</a>. Also, you can contact the Joint Chinese University of Hong Kong- New Territories East Cluster Clinical Research Ethics Committee. Tel. no.: 3505 3935.

Yours faithfully,

(Ms. CHEUNG JANICE)

Version no. 2 08/08/2022

| <b>Statement of Consent</b> | Code: |
|---|---|
| I (Name in English) carried out by Cheung Janice with a topic title program on the mental health literacy of nurs controlled trial". | |
| I confirmed that I have read the information any questions I asked. I understood the nature information collected will be kept by the resestudy. | e of this study and agree that the |
| I understand there are no known risks or<br>participation. I have had the opportunity to as<br>questions that I have asked to have been answ<br>that my participation is voluntary and confide<br>the study at any time without giving a reason. | sk questions about the study and any vered to my satisfaction. I understand ential. I have the right to withdraw from |
| By signing below, I indicate my consent to: | |
| ☐ Take part in the study. | |
| Signature of participant | Signature of the person obtaining consent |
| Name of participant | Name of the person obtaining consent |
| (Preferable Gmai | 1) |
| Email addres | SS |
| Telephon | ne |
| Dat | te Date |